CLINICAL TRIAL: NCT01923727
Title: A Phase I/IIA Study of PET Imaging With 89Zr-Df-IAb2M in Patients With Metastatic Prostate Cancer
Brief Title: Phase I/IIA Study of PET Imaging With 89Zr-Df-IAB2M in Metastatic Prostate Cancer
Acronym: IAB2M
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 002-2012
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2016-08

CONDITIONS: Metastatic Prostate Cancer
Keywords: [89Zr]Df-IAB2M; Prostate; PET Scan
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 89Zr-Df-IAB2M

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [89Zr]Df-IAB2M (Experimental): A single intravenous infusion of 5 mCi of [89Zr]Df-IAB2M in mass doses of either 10 mg, 20 mg or 50 mg (optional).
  Interventions: Biological: [89Zr]Df-IAB2M

INTERVENTIONS:
Biological: [89Zr]Df-IAB2M — A single intravenous infusion of 5 mCi of [89Zr]Df-IAB2M in a mass dose of 10 mg, 20mg or 50mg.

SUMMARY:
This is a Phase I/IIa study evaluating the safety and feasibility of [89Zr]Df-IAB2M as an immunoPET tracer for metastatic prostate cancer. Individuals participating in this study will have a FDG PET scan, as well as four (4) PET scans (over a 3 day period) following the injection of [89Zr]Df-IAB2M PET tracer. Three different dosing levels will be explored. The purpose of the study is to demonstrate the safety of [89Zr]Df-IAB2M, ability to detect prostate cancer, and optimal time point and dose level for imaging.

DETAILED DESCRIPTION:
IAB2M is an approximately 80 kDA molecular weight antibody fragment (a "Minibody"). Limited (Phase 0/Proof-of-concept) patient experience with this biologic targeting agent has been previously obtained with SPECT imaging Ex-US, demonstrating targeting of soft tissue and bone lesions in advanced metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult male >/= 18 years of age
* Patients with histologically confirmed prostate cancer
* Progressive disease manifest (within 6 weeks of screening) by either

  * imaging modalities (bone scan, MRI or CT) OR
  * biochemical progression (PSA)
* Performance status of 60 or higher on Karnofsky scale
* Subject's schedule permits compliance with all study procedures
* Ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* Previous anaphylactic reaction to huJ591 antibody or FDG imaging
* On any new anticancer therapy (GnRH analog allowed) while on the study
* Hepatic lab values: Bilirubin>1.5 ULN; AST/ALT >2.5 ULN; Albumin < 2 g/dL; GGT > 2.5 ULN if Alkaline Phostphatase >2.5 ULN
* Renal lab values: Creatinine > 1.5 ULN
* Other severe acute or chronic medical condition that may increase the risk associated with study participation or investigational product administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety of [89Zr]Df-IAB2M PET in patients with metastatic prostate cancer. | Day 1 (Infusion Day) through Day 7
  To assess the safety of a single dose of of [89Zr]Df-IAB2M

SECONDARY OUTCOMES:
[89Zr]Dr-IAB2M PET/CT quantitative assessment of metastatic prostate cancer | Day 1 (Infusion Day) to Day 3
  To determine the ability of 89Zr-Df-IAb2M PET to detect known sites of disease in patients with metastatic prostate cancer
Optimal parameters for imaging with [89Zr]Df-IAB2M | Day 1 (Infusion Day) to Day 3
  To evaluate the mass dose and hours post infusion that provides optimal detection of metastatic prostate cancer
Sensitivity of [89Zr]Df-IAB2M to detect metastatic prostate cancer | Up to 4 weeks
  To compare the results of the biopsy and FDG PET scan to the [89Zr]Df-IAB2M images

OTHER OUTCOMES:
Determine the radiation dose levels from a single infusion of [89Zr]Df-IAB2M in individuals with metastatic prostate cancer | Day 1 (Infusion Visit) to Day 3
  Evaluate the biodistribution of [89Zr]Df-IAB2M with PET/CT scans, whole body counts and blood samples to determine the radiation dose to organs in individuals with metastatic prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes